CLINICAL TRIAL: NCT06865781
Title: Minimizing Overnight Vital Signs to Improve Sleep in Hospitalized Children
Brief Title: Vital Signs Reduction Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1052853
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hospitalization
Keywords: pediatric; hospitalization; vital signs; sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Receive standard of care vital signs
- Intervention group (Experimental): Will not receive vital signs at 0000 or 0400 of study night.
  Interventions: Other: Forgone overnight vital signs

INTERVENTIONS:
Other: Forgone overnight vital signs — No vital signs (temp, heart rate, respiratory rate, blood pressure, oxygen saturation) taken at 0000 or 0400
  Arms: Intervention group

SUMMARY:
Overnight vital signs are typically done every four hours on pediatric acute care units, despite limited evidence supporting the efficacy of this practice. Additionally, vital signs are often ordered and collected without considering the patient's clinical status or the potential impact that they may have on sleep. The purpose of this study is to understand the effect of forgone overnight vital signs on sleep quality and duration among children hospitalized in medical-surgical units, compared with children who receive standard of care vital signs.

DETAILED DESCRIPTION:
Patients will be screened at Primary Children's Hospital. Patients who are deemed eligible to forgo overnight vital signs will be considered for study. After written informed consent (parental permission/assent) is obtained, subjects who meet eligibility criteria will be allocated 1:1 to 2 treatment arms in sequential order: Group 1: standard of care vital signs monitoring and Group 2: no overnight vital signs at 0000 and 0400. The study period is approximately 24 hours, including one night of sleep. All participants will wear an actigraphy watch for one night and complete a sleep diary and sleep disruption survey after the study night. The primary endpoint is total sleep time, as measured by actigraphy. Secondary endpoints include nocturnal wake frequency, nocturnal wake duration (actigraphy), self-reported total sleep time (sleep diary), self-reported overnight disruptions (sleep diary), self-reported restfulness upon waking (sleep diary), self-reported sleep disturbances (sleep disturbance survey).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at Primary Children's Hospital on units 3 Southeast, 3 Northeast, 3 Northwest
* Age 1-18 years
* Pediatric Early Warning Score ≤ 1 at 2000
* A parent/home caregiver present to consent to study
* Patient and home caregiver speak English or Spanish.
* Deemed appropriate for forgone overnight vital signs by care team (attending MD/Advanced Practice Provider and bedside RN).

Exclusion Criteria:

* Pre-existing diagnosis of hypertension, kidney disease, pulmonary hypertension, chronic lung disease, congenital heart disease causing cardiopulmonary compromise, obstructive sleep apnea, seizure disorder, neuromuscular disability.
* Patients requiring O2 monitoring at home.
* The following medications in the previous 24 hours: opioids, intravenous immunoglobulin, intravenous magnesium, continuous albuterol, benzodiazepines, other sedating medications beyond home regimen.
* Anaphylaxis within 24 hours
* Within the first 24 hours post-operative period
* Requiring oxygen above baseline
* Fever in the last 24 hours.
* Sepsis alert in the last 72 hours.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Total sleep time | From enrollment to end of treatment at 24 hours
  Measured by actigraphy

SECONDARY OUTCOMES:
Nocturnal wake frequency | From enrollment to the end of treatment at 24 hours
  By actigraphy
Nocturnal wake duration | From enrollment to the end of treatment at 24 hours
  By actigraphy
Total sleep time | From enrollment to the end of treatment at 24 hours
  By self report via sleep diary
Overnight disruptions | From enrollment to the end of treatment at 24 hours
  By self report via sleep diary
Restfulness upon waking | From enrollment to the end of treatment at 24 hours
  By self report via sleep diary
Sleep disturbances | From enrollment to the end of treatment at 24 hours
  By self report via Patient-Reported Outcomes Measurement Information System (PROMIS) sleep disturbance survey

CONTACTS AND LOCATIONS:
Overall Officials: Leandra Bitterfeld, MSN, Principal Investigator — Intermountain Primary Children's Hospital
Locations (1):
- Intermountain Primary Children's Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared because participant consent does not include data sharing outside of the study team.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT06865781/Prot_SAP_000.pdf